CLINICAL TRIAL: NCT02751151
Title: Photodynamic Therapy for Prevention of Nonmelanoma Skin Cancer in Organ Transplant Recipients
Acronym: PDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-1845
Record Dates: First submitted 2016-03-21; First posted 2016-04-26 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Nonmelanoma Skin Cancers
MeSH Terms: interventions — Aminolevulinic Acid; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Levulan Kerastick (aminolevulinic acid) solution applied to the face and/or scalp (if both are needed, treated separately on back to back days); with an incubation period of 2.5 hours. Blue light photodynamic therapy utilizing the DUSA BLU-U device, illumination: 1000 seconds (16 min, 40 secs), will be administered
  Interventions: Other: have Levulan Kerastick (aminolevulinic acid) solution

INTERVENTIONS:
Other: have Levulan Kerastick (aminolevulinic acid) solution — Levulan Kerastick (aminolevulinic acid) solution applied to the face and/or scalp (if both are needed, treated separately on back to back days); with an incubation period of 2.5 hours. Blue light photodynamic therapy utilizing the DUSA BLU-U device, illumination: 1000 seconds (16 min, 40 secs), will be administered

SUMMARY:
The study will draw patients from the Transplant Dermatology specialty clinic, where the investigators see organ transplant recipients (OTR) for regular screening and serve as a regional referral center for this population. Enrollment will be limited to 20 patients. Inclusion criteria are organ transplant recipients status, active immunosuppression for at least 5 years, and history of at least one NMSC.

DETAILED DESCRIPTION:
Patients will receive Levulan Kerastick (aminolevulinic acid) to the face and/or scalp (if both are needed, treated separately on back to back days); incubation: 2.5 hours and blue light photodynamic therapy utilizing the DUSA BLU-U device; illumination: 1000 seconds (16 min, 40 secs); administered quarterly for 3 years. Patients who change systemic immunosuppression regimens or add or increase systemic chemoprevention while in the study will be excluded from the overall analysis. The patients will be evaluated by the principal investigator every 3 months, prior to photodynamic therapy (PDT) administration.

Primary endpoints include:

1. development of non melanoma skin cancers (NMSC) lesions and
2. assessment of actinic damage score.

The primary endpoint will be development of new skin cancers at 3 years, based on comparison to rate at baseline from previous (x) year(s) using absolute slope value for number prior to treatment vs. number after treatment. The patients will serve as their own controls and the investigators will analyze the delta in development of non melanoma skin cancers and actinic damage score pre- and post- treatment.

Additionally, an actinic damage score will be assigned based on the number of actinic keratosis on initial evaluation. At each 3 month follow up visit, the actinic damage score will be reassessed. The investigators will be able to secondarily analyze the delta in the actinic damage score on treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has been the recipient of any solid organ transplant.
2. Active immunosuppression for at least 5 years
3. History of at least one NMSC
4. Subject is willing to sign an informed consent to participate in this study.

Exclusion Criteria:

1. Patient is not appropriate candidate for treatment or research trial per treating physician
2. Patient has a mental health condition that makes them unable to participate in this research trial, per PI judgment.
3. Patient is on additional immunosuppression for diagnosis unrelated to organ transplant -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Number of non melanoma skin cancers in organ transplant recipients | through study completion, an average of 2 years

SECONDARY OUTCOMES:
Reduction of actinic keratosis damage/epidermal dysplasia in organ transplant recipients as assessed by physician and graded per actinic damage scale | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer DeSimone, MD, Principal Investigator — Physician
Locations (1):
- Inova Melanoma Na Skin Oncology Center, Fairfax, Virginia, United States